CLINICAL TRIAL: NCT07059273
Title: An Observational, Prospective, Real-world Data Registry in Chronic Obstructive Pulmonary Disease (COPD) Patients Suffering From Frequent Exacerbations (AIREIC)
Brief Title: A COPD Data Registry for Participants With Frequent Exacerbations
Acronym: AIREIC
Status: Not yet recruiting | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: BA45495
Record Dates: First submitted 2025-06-24; First posted 2025-07-10 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD Arm: Participants with COPD with frequent exacerbations will be followed from the date of enrollment until death, loss to follow up, withdrawal of consent, or the end of the follow-up period, for up to 3 years.

SUMMARY:
This registry will collect data on COPD, including the course of disease, treatment patterns, and potential new therapies. The registry will also track the experience of participants and caregivers in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD for at least 12 months
* On stable, standard of care (SoC) COPD maintenance therapy
* Have experienced at least 2 exacerbations (moderate or severe) in the last 12 months, with one of them occurring while on SoC therapy

Exclusion Criteria:

* In palliative treatment
* Participating in any interventional drug trials

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants at least 40 years of age that have had a COPD diagnosis for at least 12 months, are on stable maintenance therapy, and who have experienced at least two exacerbations in the last 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2026-05-18 (Estimated); Primary Completion 2030-11-18 (Estimated); Study Completion 2030-11-18 (Estimated)

PRIMARY OUTCOMES:
Disease course of participants enrolled in COPD registry | Up to 3 years
Treatment patterns of participants enrolled in COPD registry | Up to 3 years
  Treatment patterns of participants enrolled in COPD registry would be monitored through medical records and the changes in the standard of care and potentially moving to other treatments such as biologics.
Number of novel therapies for participants enrolled in COPD registry | Up to 3 years
  Through medical records, the number and type of novel therapies would be assessed for participants enrolled in COPD registry.
Health care utilization (HCU) by participants enrolled in COPD registry as measured by number of medical visits | Up to 3 years
HCU by participants enrolled in COPD registry as measured by types of medical care institutions visited | Up to 3 years
Quality of life (QoL) of participants enrolled in COPD registry as measured by the Chronic Airways Assessment Test (CAAT) | Up to 3 years
QoL of participants enrolled in COPD registry as measured by the EQ-5D Five Levels plus respiratory dimension (EQ-5D-5L+R) questionnaire | Up to 3 years
QoL of participants enrolled in COPD registry as measured by the Work Productivity and Impairment (WPAI)-COPD | Up to 3 years
QoL of participants enrolled in COPD registry as measured by the COPD treatment satisfaction questionnaire | Up to 3 years
QoL of participants enrolled in COPD registry as measured by the exacerbation experience questionnaire | Up to 3 years
Caregiver burden as measured by the Zarit Burden Interview 12-item (ZBI-12) | Up to 3 years
Caregiver burden as measured by the Work Productivity and Impairment (WPAI) questionnaire | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche

IPD SHARING:
Plan to Share IPD: No